CLINICAL TRIAL: NCT02052310
Title: A Phase 3, Multicenter, Randomized, Open-Label, Active-Controlled Study of the Efficacy and Safety of FG-4592 in the Treatment of Anemia in Incident-Dialysis Patients
Brief Title: Safety and Efficacy Study of Roxadustat (FG-4592) for the Treatment of Anemia in End-Stage Renal Disease (ESRD) Newly Initiated Dialysis Participants
Acronym: Himalayas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-063; 2013-002753-30 (EudraCT Number)
Record Dates: First submitted 2014-01-06; First posted 2014-02-03 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Anemia in Incident Dialysis Patients
Keywords: Anemia; Chronic Kidney Disease; Hemoglobin; End-Stage Renal Disease; Incident-Dialysis; Erythropoieitin; Erythropoieisis stimulating-agent; Roxadustat; AZD9941; ASP1517; FG4592
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — roxadustat; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Participants will receive roxadustat tablets, administered orally 3 times weekly (TIW). Initial roxadustat dose will be based on a tiered, weight-based dosing scheme (low weight [≤70 kilograms (kg)] and high weight [>70 to 160 kg] participants will receive 70 and 100 milligrams [mg] roxadustat, respectively). Dose adjustment to achieve correction and subsequent maintenance of target hemoglobin (Hb) values (10-12 grams [g]/deciliter [dL]) will be based upon regular monitoring of Hb. The maximum roxadustat dose is 3.0 mg/kg per dose or 400 mg per administration (whichever is lower).
  Interventions: Drug: Roxadustat
- Epoetin Alfa (Active Comparator): Participants on hemodialysis (HD) will receive epoetin alfa, administered intravenously (IV) TIW, with starting doses and dose adjustment rules as per United States Package Insert (USPI) or summary of product characteristics (SmPC). Participants on home HD or peritoneal dialysis (PD) will receive epoetin alfa, administered subcutaneously (SC) as per the country-specific product label (USPI or SmPC) or local standard of care (SOC).
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be administered per dose and schedule specified in the arm.
  Other Names: ASP1517; AZD9941; FG-4592
  Arms: Roxadustat
Drug: Epoetin Alfa — Epoetin alfa will be administered TIW according to the epoetin alfa USPI or SmPC, or local SOC.
  Other Names: Procrit; Epogen
  Arms: Epoetin Alfa

SUMMARY:
The purpose of this study is to determine whether roxadustat is safe and effective in the treatment of anemia in participants who have just begun dialysis treatment for ESRD.

DETAILED DESCRIPTION:
There is a screening period of up to 6 weeks, a treatment period of a minimum of 52 weeks and a maximum of approximately up to 3 years after last participant is randomized, and a post-treatment follow-up period of 4 weeks. Participants will be randomized in a 1:1 ratio to receive either open-label roxadustat or epoetin alfa (active control).

ELIGIBILITY:
Inclusion Criteria:

* Participant has been informed of the investigational nature of this study and has given written informed consent in accordance with institutional, local, and national guidelines.
* Receiving HD or PD for ESRD for a minimum of 2 weeks and a maximum of 4 months, prior to randomization.
* Hemodialysis access consisting of an arteriovenous (AV) fistula, AV graft, or tunnelled (permanent) catheter; or PD catheter in use.
* Mean of the two most recent predialysis Hb values during the Screening Period, obtained at least 2 days apart, must be ≤ 10.0 g/dL, with a difference of ≤ 1.3 g/dL between the highest and the lowest values. The last Hb value must be drawn within 10 days prior to randomization.
* Ferritin ≥ 100 nanograms (ng)/milliliter (mL) (≥ 220 picomoles (pmol)/L); participants with ferritin level < 100 ng/mL(<220 pmol/L) during screening, qualify after receiving iron supplement (per local standard of care), without the need to retest ferritin prior to randomization.
* Transferrin saturation ≥ 20%; participants with TSAT level < 20% during screening, qualify after receiving iron supplement (per local standard of care), without the need to retest TSAT prior to randomization.
* Serum folate level, performed within 8 weeks prior to randomization ≥ lower limit of normal (LLN); participants with serum folate level < LLN during screening, qualify after receiving folate supplement (per local standard of care), without the need to retest folate prior to randomization.
* Serum vitamin B12 level, performed within 8 weeks prior to randomization ≥ LLN; participants with vitamin B12 level < LLN during screening, qualify after receiving B12 supplement (per local standard of care), without the need to retest B12 prior to randomization.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3 * upper limit of normal (ULN), and total bilirubin ≤ 1.5 * ULN.
* Body weight up to 160 kg (HD participants: dry weight).

Exclusion Criteria:

* Total duration of prior effective ESA use must be ≤3 weeks within the preceding 12 weeks at the time informed consent is obtained.

Specific dosing guidance, depending on the type of ESAs, injected IV or SC within 12 weeks prior to start of screening are as follows:

i) Short-acting ESAs (EPO-alfa or equivalents) - IV: Up to 9 doses, last EPO dose must be ≥2 days prior to start of screening; SC: Up to 3 doses, last EPO dose must be ≥1 week (7 days) prior to start of screening ii) Darbepoetin - IV: Up to 3 doses, last darbepoetin dose must be ≥1 week (7 days) prior to start of screening; SC: Up to 2 doses, last darbepoetin dose must be ≥2 weeks (14 days) prior to start of screening iii) Continuous erythropoietin receptor activator (CERA) IV and SC: Up to 2 doses; last CERA dose must be ≥2 weeks (14 days) prior to start of screening

* Intravenous iron: there is no restriction regarding IV iron use during screening, provided it is administered in accordance with local SOC.
* Red blood cell transfusion within 4 weeks prior to randomization.
* Active, clinically significant infection that could be manifested by white blood cell (WBC) count > ULN, and/or fever, in conjunction with clinical signs or symptoms of infection at the time of randomization.
* History of chronic liver disease (for example, chronic infectious hepatitis, chronic auto-immune liver disease, cirrhosis, or fibrosis of the liver).
* New York Heart Association Class III or IV congestive heart failure at screening.
* Myocardial infarction, acute coronary syndrome, stroke, seizure, or a thromboembolic event within a major vessel (excluding vascular dialysis access) (for example, deep vein thrombosis or pulmonary embolism) within 12 weeks prior to randomization.
* Uncontrolled hypertension, in the opinion of the Investigator, (for example, that requires a change in anti-hypertensive medication) within 2 weeks prior to randomization.
* Renal imaging performed within 12 weeks prior to randomization indicative of a diagnosis or suspicion (for example, complex kidney cyst of Bosniak Category 2 or higher) of renal cell carcinoma.
* History of malignancy, except for the following: cancers determined to be cured or in remission for ≥ 5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps.
* Positive for any of the following: human immunodeficiency virus (HIV); hepatitis B surface antigen (HBsAg); or anti-hepatitis C virus antibody (anti-HCV Ab).
* Chronic inflammatory disease that could impact erythropoiesis (for example, systemic lupus erythematosus, rheumatoid arthritis, celiac disease) even if it is currently in remission.
* Known, untreated proliferative diabetic retinopathy, diabetic macular edema, macular degeneration, or retinal vein occlusion (participants who are already blind for the above reasons qualify to participate).
* Known history of myelodysplastic syndrome or multiple myeloma.
* Known hereditary hematologic disease such as thalassemia or sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than chronic kidney disease (CKD).
* Known hemosiderosis, hemochromatosis, coagulation disorder, or a hypercoagulable condition.
* Organ transplant: participants with any of the following:

  1. Experienced rejection of a transplanted organ within 6 months of transplantation
  2. Currently on high doses of immunosuppressive therapy (per discretion of the Investigator)
  3. Scheduled for organ transplantation. Note: being on a waiting list for kidney transplant is not exclusionary
* Anticipated elective surgery, except for vascular access surgery or dialysis catheter placement, that is expected to lead to significant blood loss, or anticipated elective coronary revascularization.
* Active or chronic gastrointestinal bleeding.
* Any prior treatment with roxadustat or a hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI).
* Use of iron-chelating agents within 4 weeks prior to randomization.
* Known hypersensitivity reaction to any ESA.
* Use of an investigational drug or treatment, participation in an investigational study, or presence of an expected carryover effect of an investigational treatment, within 4 weeks prior to randomization.
* Anticipated use of dapsone or androgens at any dose amount or chronic use of acetaminophen or paracetamol > 2.0 g/day during the study.
* History of alcohol or drug abuse within 6 months prior to randomization.
* Females of childbearing potential, unless using contraception as detailed in the protocol; male participants with sexual partners of childbearing potential who are not on birth control unless the male participant agrees to use contraception.
* Pregnant or breastfeeding females.
* Any medical condition that, in the opinion of the Investigator, may pose a safety risk to a participant in this study, may confound efficacy or safety assessment, or may interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bradley, PhD, Study Director — Kyntra Bio
Locations (98):
- United States (28):
  - Investigational Site, Chula Vista, California
  - Investigational Site, La Mesa, California
  - Investigational Site, San Diego, California
  - Investigational Site, Coral Springs, Florida
  - Investigational Site, Lauderdale Lakes, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Tampa, Florida
  - Meridian, Meridian, Idaho
  - Investigational Site, Shreveport, Louisiana
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Pontiac, Michigan
  - Investigational Site, Brookhaven, Mississippi
  - Investigational Site, Columbus, Mississippi
  - Investigational Site, Gulfport, Mississippi
  - Investigational Site, Tupelo, Mississippi
  - Investigational Site, Saint Ann, Missouri
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Portsmouth, New Hampshire
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, Durham, North Carolina
  - Investigational Site, New Bern, North Carolina
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Columbia, South Carolina
  - Investigational Site, Orangeburg, South Carolina
  - Investigational Site, Sumter, South Carolina
  - Investigational Site, Knoxville, Tennessee
  - Investigational Site, Edinburg, Texas
  - Investigational Site, Houston, Texas
- Argentina (2):
  - Investigational Site, Serandi, Buenos Aires
  - Investigational Site, Santa Fe, IX Region
- Bulgaria (11):
  - Investigational Site, Burgas
  - Investigational site, Dobrich
  - Investigational site, Pazardzhik
  - Investigational site, Pernik
  - Investigational Site, Pleven
  - Investigational Site, Plovdiv
  - Investigational site, Rousse
  - Investigational Site, Sofia
  - Investigational site, Sofia
  - Invesigational Site, Stara Zagora
  - Investigational Site, Varna
- Chile (2):
  - Investigational Site, La Serena, Coquimbo Region
  - Investigational Site, Temuco, Región de la Araucanía
- Colombia (2):
  - Investigational Site, Barranquilla, Atlántico
  - Investigational Site, Barranquilla
- Latvia (3):
  - Investigational Site, Riga
  - Invetigational Site, Riga
  - Investigational Site, Ventspils
- Malaysia (5):
  - Investigational Site, Miri, Sarawak
  - Investigational Site, Alor Star
  - Investigational Site, George Town
  - Investigational Site, Kuala Lumpur
  - Investigational Site, Taiping
- Mexico (2):
  - Investigational Site, Aguascalientes
  - Investigational Site, San Luis Potosí City
- Poland (5):
  - Investigational Site, Chorzów
  - Investigational Site, Golub-Dobrzyń
  - Investigational Site, Inowrocław
  - Investigational Site, Katowice
  - Investigational Drug, Pruszków
- Romania (5):
  - Investigational Site, Bucharest, District 3
  - Investigational Site, Bucharest
  - Investigational Site, Craiova
  - Investigational Site, Slatina
  - Investigational Site, Târgu Mureş
- Russia (17):
  - Investigational Site, Kaluga, Russian Federation
  - Investigational Site, Krasnodar, Russian Federation
  - Investigational Site, Moscow, Russian Federation
  - Investigational Site, Nizhny Novgorod, Russian Federation
  - Investigational Site, Petrozavodsk, Russian Federation
  - Investigational Site, Saint Petersburg, Russian Federation
  - Investigational Site, Smolensk, Russian Federation
  - Investigational Site, Moscow, Russian Ferderation
  - Investigational Site, Kolomna
  - Investigational Site, Krasnodar
  - investigational Site, Moscow
  - Investigational Site, Novorossiysk
  - Investigational site, Omsk
  - Investigational Site, Orenburg
  - Investigational Site, Rostov-on-Don
  - Investigational Site, Saint Petersburg
  - Investigational site, Saint Petersburg
- South Korea (5):
  - Investigational site, Goyang-si, Gyeonggi-do
  - Investigational Site, Guri-si, Gyeonggi-do
  - Investigational Site, Seongnam-si, Gyeonggi-do
  - Investigational Site, Anyang-si
  - Investigational Site, Seoul
- Taiwan (3):
  - Investigational Site, Kaohsiung City
  - Investigational Site,, New Taipei City
  - Investigational Site, Taichung
- Thailand (2):
  - Investigational Site, Bangkok
  - Investigational Site, Chiang Mai
- Ukraine (6):
  - Investigational Site, Ivano, Frankivisk
  - Investigational Site, Karkiev
  - Investigational Site, Kiev
  - Investigational Site, Mykolayiv
  - Investigational Site, Ternopil
  - Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Martin S, Jiletcovici A, Dellanna F, Akizawa T, Barratt J. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Four Global Roxadustat Phase 3 Trials. Adv Ther. 2024 Apr;41(4):1553-1575. doi: 10.1007/s12325-023-02728-2. Epub 2024 Feb 16. PMID 38363466
- [Derived] Barratt J, Dellanna F, Portoles J, Choukroun G, De Nicola L, Young J, Dimkovic N, Reusch M. Safety of Roxadustat Versus Erythropoiesis-Stimulating Agents in Patients with Anemia of Non-dialysis-Dependent or Incident-to-Dialysis Chronic Kidney Disease: Pooled Analysis of Four Phase 3 Studies. Adv Ther. 2023 Apr;40(4):1546-1559. doi: 10.1007/s12325-023-02433-0. Epub 2023 Feb 7. PMID 36749544
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either roxadustat or epoetin alfa.
Groups:
- Roxadustat: Participants received roxadustat tablets, administered orally 3 times weekly (TIW). Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low weight [≤70 kilograms (kg)] and high weight [>70 to 160 kg] participants received 70 and 100 milligrams [mg] roxadustat, respectively). Dose adjustment to achieve correction and subsequent maintenance of target hemoglobin (Hb) values (10-12 grams [g]/deciliter [dL]) was based upon regular monitoring of Hb. The maximum roxadustat dose was 3.0 mg/kg per dose or 400 mg per administration (whichever was lower). The maximum treatment duration was 227.9 weeks.
- Epoetin Alfa: Participants on hemodialysis (HD) received epoetin alfa, administered intravenously (IV) TIW, with starting doses and dose adjustment rules as per United States Package Insert (USPI) or summary of product characteristics (SmPC). Participants on home HD or peritoneal dialysis (PD) received epoetin alfa, administered subcutaneously (SC) as per the country-specific product label (USPI or SmPC) or local standard of care (SOC). The maximum treatment duration was 226.9 weeks.
Period: Overall Study
Arm/Group | Roxadustat | Epoetin Alfa
Started | 522 | 521
Received at Least 1 Dose of Study Drug | 522 | 517
Completed | 307 | 309
Not Completed | 215 | 212
Not completed — Death | 64 | 54
Not completed — Withdrawal by Subject | 37 | 49
Not completed — Other than specified | 32 | 29
Not completed — Adverse Event | 29 | 22
Not completed — Kidney Transplant | 23 | 29
Not completed — Physician Decision | 14 | 7
Not completed — Lack of Efficacy | 6 | 1
Not completed — Site Terminated by Sponsor | 5 | 13
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 1 | 6

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population included all randomized participants.
Groups:
- Roxadustat: Participants received roxadustat tablets, administered orally TIW. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low weight [≤70 kg] and high weight [>70 to 160 kg] participants received 70 and 100 mg roxadustat, respectively). Dose adjustment to achieve correction and subsequent maintenance of target Hb values (10-12 g/dL) was based upon regular monitoring of Hb. The maximum roxadustat dose was 3.0 mg/kg per dose or 400 mg per administration (whichever was lower). The maximum treatment duration was 227.9 weeks.
- Epoetin Alfa: Participants on HD received epoetin alfa, administered IV TIW, with starting doses and dose adjustment rules as per USPI or SmPC. Participants on home HD or PD received epoetin alfa, administered SC as per the country-specific product label (USPI or SmPC) or local SOC. The maximum treatment duration was 226.9 weeks.
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Epoetin Alfa | Total
Number analyzed (Participants) | 522 | 521 | 1043
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 381 | 391 | 772
  >=65 years | 141 | 130 | 271
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 214 | 427
  Male | 309 | 307 | 616
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 77 | 176
  Not Hispanic or Latino | 423 | 444 | 867
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 415 | 400 | 815
  Race: Black/African American | 44 | 50 | 94
  Race: Asian | 43 | 51 | 94
  Race: Other | 19 | 16 | 35
  Race: American Indian/ Alaskan Native | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: US (FDA) Submission: Mean Hb Change From Baseline to The Average Level During The Evaluation Period (Week 28 to Week 52), Regardless of Rescue Therapy (ITT Population)
Description: Hb values under the influence of rescue therapy were not censored for the primary analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (erythropoiesis-stimulating agent [ESA]) or red blood cell (RBC) transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment. The intermittent missing Hb data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the Monte Carlo Markov Chain (MCMC) imputation model, Monotone missing data were imputed by regression from its own treatment group.
Time Frame: Baseline (Day 1, Week 0), Week 28 to 52
Population: The ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 521
g/dL
  Baseline | 8.43 (1.044) | 8.46 (0.964)
  Change at Week 28 to 52 | 2.57 (1.269) | 2.36 (1.214)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using the multiple imputation (MI) strategy by combining the results of analysis of covariance (ANCOVA) model with baseline Hb as a covariate, and treatment, region and cardiovascular/cerebrovascular/thromboembolic medical history (yes vs. no) as factors; Test type: Non-Inferiority — Non-inferiority was established if the 2-sided 95% confidence interval (CI) for the treatment difference in least square (LS) means from MI ANCOVA model between the 2 treatment groups lay entirely above -0.75 g/dL; p = 0.0005, ANCOVA; ANCOVA with multiple imputation; LS Mean Difference = 0.18, 95% CI 2-sided [0.079 to 0.287], Standard Error of Mean 0.053

2. Primary Outcome: Ex-U.S. Submission: Hb Responder Rate- Percentage of Participants Who Achieved a Hb Response at 2 Consecutive Visits at Least 5 Days Apart During First 24 Weeks of Treatment, Without Rescue Therapy Within 6 Weeks Prior to the Hb Response (PPS Population)
Description: Hb response was defined, using central laboratory values, as: Hb ≥11.0 g/dL and a Hb increase from baseline by ≥1.0 g/dL in participants whose baseline Hb >8.0 g/dL, or increase in Hb ≥2.0 g/dL in participants whose baseline Hb ≤8.0 g/dL. Rescue therapy for roxadustat treated participant was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion.
Time Frame: Baseline (Day 1, Week 0) up to Week 24
Population: The per protocol set (PPS) population included all participants in the full analysis set (FAS) population (all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment) who received at least 8 weeks of treatment and were without major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 490 | 468
percentage of participants | 88.2 | 84.4
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; For the difference of responder rates between 2 treatment groups, the CI was analyzed from the Miettinen & Nurminen approach adjusting for randomization stratification factors; Test type: Non-Inferiority — Non-inferiority was established if the lower bound of the 2-sided 95% CI for the treatment difference for the responder rates (roxadustat minus epoetin alfa) calculated based on the Miettinen & Nurminen approach, adjusting for stratification factors, was greater than -15%; Responder Rate Difference = 3.5, 95% CI 2-sided [-0.7 to 7.7]

3. Secondary Outcome: US (FDA Submission): Hb Responder Rate- Percentage of Participants Who Achieved a Hb Response at 2 Consecutive Visits at Least 5 Days Apart During First 24 Weeks of Treatment, Without Rescue Therapy Within 6 Weeks Prior to the Hb Response (ITT Population)
Description: as for outcome 2
Time Frame: Baseline (Day 1, Week 0) up to Week 24
Population: The ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 521
percentage of participants | 84.3 | 79.5
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; For the difference of responder rates between 2 treatment groups, the CI analyzed was from the Miettinen & Nurminen approach adjusting for randomization stratification factors; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Responder Rate Difference = 4.3, 95% CI 2-sided [-0.1 to 8.7]

4. Secondary Outcome: Ex-US Submission: Mean Hb Change From Baseline to The Average Level During The Evaluation Period (Week 28 to Week 52), Regardless of Rescue Therapy (PPS Population)
Description: Hb values under the influence of rescue therapy were censored up to 6 weeks in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment. The intermittent missing Hb data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the MCMC imputation model, Monotone missing data were imputed by regression from its own treatment group.
Time Frame: Baseline (Day 1, Week 0), Week 28 to 52
Population: The PPS population included all participants in the FAS population (all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment) who received at least 8 weeks of treatment and were without major protocol violations. Here, 'Number analyzed' signifies participants with non-missing data for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 490 | 468
g/dL
  Baseline | 8.43 (1.043) | 8.43 (0.963)
  Change at Week 28 to 52: number analyzed (Participants) | 434 | 419
  Change at Week 28 to 52 | 2.62 (1.292) | 2.44 (1.209)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using mixed model for repeated measures (MMRM) with baseline Hb as a covariate, and treatment, visit, visit-by-treatment interaction and randomization stratification factors except mean qualifying screening hemoglobin (≤8.0 vs. >8.0 g/dL) as fixed effects; Test type: Non-Inferiority — Non-inferiority was established if the 2-sided 95% CI for the treatment difference in LS means of change from baseline Hb averaged over Weeks 28 to 52 lay entirely above -0.75 g/dL; p = 0.0148, Mixed Models Analysis; LS Mean Difference = 0.16, 95% CI 2-sided [0.032 to 0.296], Standard Error of Mean 0.067

5. Secondary Outcome: Mean Change From Baseline in Low-Density Lipoprotein (LDL) Cholesterol Averaged Over Weeks 12 to 24
Description: Baseline LDL Cholesterol was defined as the mean of values obtained within 6 weeks prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Week 12 to 24
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment. Here, 'Number analyzed' signifies participants with non-missing data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 513
mg/dL
  Baseline | 109.12 (38.833) | 109.22 (35.914)
  Change at Weeks 12 to 24: number analyzed (Participants) | 487 | 481
  Change at Weeks 12 to 24 | -23.80 (29.996) | -5.39 (26.164)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using a MMRM with baseline LDL cholesterol as a covariate, and treatment, visit, visit-by-treatment interaction and randomization stratification factors as fixed effects; Test type: Superiority — Superiority was declared if the upper bound of the 2-sided 95% CI of the difference between roxadustat and epoetin alfa (roxadustat - epoetin alpha) was less than 0; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -18.34, 95% CI 2-sided [-21.448 to -15.232], Standard Error of Mean 1.584

6. Secondary Outcome: Mean Change From Baseline in Hb Levels Between Weeks 18 to 24 Regardless of Rescue Therapy in Participants Whose Baseline High Sensitivity C-Reactive Protein (Hs-CRP)> Upper Limit of Normal (ULN)
Description: Hb values under the influence of rescue therapy were not censored in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment. The intermittent missing Hb data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the MCMC imputation model, Monotone missing data were imputed by regression from its own treatment group.
Time Frame: Baseline (Day 1, Week 0), Week 18 to 24
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 228 | 222
g/dL
  Baseline | 8.54 (0.968) | 8.38 (0.961)
  Change at Week 18 to 24 | 2.34 (1.256) | 2.48 (1.271)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using the multiple imputation strategy by combining the results of ANCOVA model with baseline Hb as a covariate, and treatment, region and cardiovascular/cerebrovascular/thromboembolic medical history (yes vs. no) as factors; Test type: Non-Inferiority — The non-inferiority margin was fixed as a difference of -0.75; p = 0.8178, ANCOVA; ANCOVA multiple imputation; LS Mean Difference = 0.02, 95% CI 2-sided [-0.171 to 0.217], Standard Error of Mean 0.099

7. Secondary Outcome: Median Monthly IV Iron Use Per Patient-Exposure-Month (PEM) During Weeks 28 to 52
Description: Monthly iron use for each participant = Total IV iron in mg / [(last dose date - first dose date of study medication in the period)+1]/ 28.
Time Frame: Weeks 28 to 52
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/PEM
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 437 | 438
mg/PEM | 0.00 [0.0 to 1600.0] | 26.86 [0.0 to 717.7]
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using an ANCOVA model with baseline iron repletion status, treatment, and randomization stratification factors as fixed effects; Test type: Superiority; p = 0.00028, Rank ANCOVA — Threshold for significance at 0.05 level

8. Secondary Outcome: Time to First RBC Transfusion
Description: Median time to event (weeks) was calculated using Kaplan Meier Survival Estimates.
Time Frame: Baseline (Day 1, Week 0) up to last dose of study drug (maximum treatment duration was 227.9 weeks for roxadustat and 226.9 weeks for epoetin alfa)
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 513
weeks | NA [NA to NA] — Due to smaller number of participants with an event (any use of RBC transfusion), median and 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event (any use of RBC transfusion), median and 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Analysis was done using a Cox Proportional Hazards model adjusting for baseline Hb and other stratification factors except mean qualifying screening hemoglobin (<= 8.0 vs. >8.0 g/dL) as fixed effects; Test type: Non-Inferiority — The non-inferiority margin for the difference between groups was 1.8; p = 0.3284, Cox Proportional Hazards model; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.791 to 2.016]

9. Secondary Outcome: Mean Change From Baseline in Mean Arterial Pressure (MAP) Averaged Over Weeks 8 to 12
Description: Baseline MAP was defined as the last MAP value prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Weeks 8 to 12
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 521 | 513
millimeters of mercury (mmHg)
  Baseline | 99.33 (10.146) | 99.04 (9.874)
  Change at Weeks 8 to 12: number analyzed (Participants) | 494 | 494
  Change at Weeks 8 to 12 | -0.12 (8.018) | 1.15 (8.729)

10. Secondary Outcome: Time to First Exacerbation of Hypertension During Weeks 28 to 52
Description: An exacerbation of hypertension was defined as increase from baseline of ≥20 mmHg in systolic blood pressure (sBP) and sBP ≥170 mmHg or an increase from baseline of ≥15 mm Hg in diastolic blood pressure (dBP) and dBP ≥100 mmHg. Median time to event (weeks) was calculated using Kaplan Meier Survival Estimates.
Time Frame: Weeks 28 to 52
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 513
weeks | NA [NA to NA] — Due to smaller number of participants with an event (exacerbation hypertension), median and 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event (exacerbation hypertension), median and 95% CI could not be calculated.

11. Secondary Outcome: Percentage of Participants With Exacerbation of Hypertension During Weeks 28 to 52
Description: Percentage of participants with exacerbation of hypertension, meeting at least one of the following criteria are reported: i) Increase in BP: An increase from baseline of ≥ 20 mmHg in sBP and sBP >170 mmHg, or an increase from baseline of ≥15 mmHg dBP and dBP >100 mmHg.
Time Frame: Weeks 28 to 52
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 513
percentage of participants | 14.0 | 15.2

12. Secondary Outcome: Time to Achieve the First Hb Response up to Week 24 Censoring for Rescue Therapy
Description: Hb values under the influence of rescue therapy were censored up to 6 weeks in the analysis. Hb response was defined, using central laboratory values, as: Hb ≥11.0 g/dL and a Hb increase from baseline by ≥1.0 g/dL in participants whose baseline Hb >8.0 g/dL, or increase in Hb ≥2.0 g/dL in participants whose baseline Hb ≤8.0 g/dL. Rescue therapy for roxadustat treated participant was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Median time to event was calculated using Kaplan Meier Survival Estimates.
Time Frame: Baseline (Day 1, Week 0) up to Week 24
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 513
weeks | 7.1 [6.1 to 8.1] | 8.1 [8.1 to 9.1]

13. Secondary Outcome: Percentage of Participants With Hb ≥10.0 g/dL Averaged Over Weeks 28 to 36 and 28 to 52, Regardless of Rescue Therapy
Description: Hb values under the influence of rescue therapy were not censored in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment.
Time Frame: Weeks 28 to 36 and 28 to 52
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 522 | 513
percentage of participants
  Weeks 28 to 36 | 73.4 | 70.8
  Weeks 28 to 52 | 73.6 | 72.5

14. Secondary Outcome: Mean Hb Change From Baseline to The Average Level During The Evaluation Period (Week 28 to Week 36), Censoring for Rescue Therapy
Description: Hb values under the influence of rescue therapy were censored up to 6 weeks in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Week 28 to 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 435 | 439
g/dL | 2.70 (1.423) | 2.46 (1.308)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1, Week 0) up to 28 days after the last dose of study drug (maximum treatment duration was 227.9 weeks for roxadustat and 226.9 weeks for epoetin alfa). Mortality presented is for the timeframe of Baseline (Day 1, Week 0) up to end of treatment (maximum treatment duration was 227.9 weeks for roxadustat and 226.9 weeks for epoetin alfa).
Description: The Safety population included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Roxadustat | Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 64/522 | 54/517
Serious Adverse Events (participants affected / at risk) | 234/522 | 218/517
Other Adverse Events (participants affected / at risk) | 291/522 | 262/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Roxadustat (N=522) | Epoetin Alfa (N=517)
Acute myocardial infarction (Cardiac disorders) | 6 | 11
Cardiac failure congestive (Cardiac disorders) | 5 | 7
Myocardial infarction (Cardiac disorders) | 5 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 5
Angina unstable (Cardiac disorders) | 3 | 5
Cardiac arrest (Cardiac disorders) | 3 | 5
Pancreatitis acute (Gastrointestinal disorders) | 5 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 | 5
Sudden Death (General disorders) | 7 | 4
Death (General disorders) | 2 | 7
Pneumonia (Infections and infestations) | 30 | 26
Peritonitis (Infections and infestations) | 12 | 12
Sepsis (Infections and infestations) | 13 | 8
Device related infection (Infections and infestations) | 9 | 3
Gangrene (Infections and infestations) | 6 | 6
Cellulitis (Infections and infestations) | 4 | 5
Device related sepsis (Infections and infestations) | 7 | 2
Septic shock (Infections and infestations) | 7 | 4
Urinary tract infection (Infections and infestations) | 6 | 4
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 39 | 21
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 5 | 2
Fluid overload (Metabolism and nutrition disorders) | 9 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 6
Ischemic stroke (Nervous system disorders) | 5 | 2
Hemorrhagic stroke (Nervous system disorders) | 3 | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Hypertensive crisis (Vascular disorders) | 9 | 12
Hypertension (Vascular disorders) | 6 | 3
Hypotension (Vascular disorders) | 7 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 2 | 1
Aortic valve disease mixed (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 3
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 3 | 2
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 4 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 4 | 4
Coronary artery insufficiency (Cardiac disorders) | 2 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Microvascular coronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 2
Cataract (Eye disorders) | 1 | 1
Diabetic ophthalmoplegia (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 1
Macular fibrosis (Eye disorders) | 0 | 1
Optic neuropathy (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastritis erosive (Gastrointestinal disorders) | 2 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 1
Complication associated with device (General disorders) | 4 | 2
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 0
Generalised oedema (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Sudden cardiac death (General disorders) | 1 | 2
Vascular stent stenosis (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Gallbladder necrosis (Hepatobiliary disorders) | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic cyst ruptured (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Porcelain gallbladder (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 3
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Corona virus infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 1
Diabetic gangrene (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Endocarditis (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Female genital tract tuberculosis (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Groin abscess (Infections and infestations) | 1 | 1
Haematoma infection (Infections and infestations) | 1 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Necrotising soft tissue infection (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 4 | 4
Osteomyelitis acute (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 3
Periumbilical abscess (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 3 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Sinusitis aspergillus (Infections and infestations) | 0 | 1
Small intestine gangrene (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 4 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Toxic shock syndrome (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 2
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 1
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 3
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1
Ischaemic neuropathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 2
Status migrainosus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Vascular encephalopathy (Nervous system disorders) | 1 | 1
Vertigo CNS origin (Nervous system disorders) | 1 | 0
Device failure (Product Issues) | 1 | 0
Device leakage (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 3 | 1
Thrombosis in device (Product Issues) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 2
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 3 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Renal papillary necrosis (Renal and urinary disorders) | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1/309 | 0/307 — This is a gender-specific AE that affects only male participants.
Scrotal oedema (Reproductive system and breast disorders) | 0/309 | 1/307 — This is a gender-specific AE that affects only male participants.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Treatment noncompliance (Social circumstances) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic rupture (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 2
Dry gangrene (Vascular disorders) | 1 | 2
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 3
Iliac artery occlusion (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2
Peripheral artery stenosis (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 1
Steal syndrome (Vascular disorders) | 1 | 1
Subgaleal haematoma (Vascular disorders) | 0 | 1
Superior vena cava stenosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
Vascular occlusion (Vascular disorders) | 1 | 0
Vascular rupture (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Vasodilatation (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Large intestinal polyp (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Ureteral necrosis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Refusal of treatment by patient (Social circumstances) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=522) | Epoetin Alfa (N=517)
Diarrhea (Gastrointestinal disorders) | 72 | 38
Nausea (Gastrointestinal disorders) | 45 | 30
Constipation (Gastrointestinal disorders) | 35 | 23
Vomiting (Gastrointestinal disorders) | 32 | 17
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 26 | 28
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 27 | 42
Procedural hypotension (Injury, poisoning and procedural complications) | 25 | 31
Hyperphosphatemia (Metabolism and nutrition disorders) | 52 | 35
Hyperkalemia (Metabolism and nutrition disorders) | 24 | 30
Muscle spasms (Musculoskeletal and connective tissue disorders) | 60 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 27
Headache (Nervous system disorders) | 57 | 43
Dizziness (Nervous system disorders) | 28 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 22
Hypertension (Vascular disorders) | 96 | 87
Hypotension (Vascular disorders) | 49 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen.

The investigator can only publish after the multisite consortium publishes (or tries to publish and fails).

FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT02052310/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02052310/SAP_001.pdf